CLINICAL TRIAL: NCT02898103
Title: Percutaneous Peripheral Nerve Stimulation (Neuromodulation) for Postoperative Analgesia: A Feasibility/Proof-of-Concept Study
Brief Title: Percutaneous Peripheral Nerve Stimulation (Neuromodulation) for Postoperative Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University California Academic Senate (Unknown); Copenhagen University Hospital at Herlev (Other); SPR Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Percutaneous PNS Postop pilot
Record Dates: First submitted 2016-09-02; First posted 2016-09-13 (Estimated); Results first posted 2021-03-15 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment group assignments were unmasked after the leads were removed 2 weeks after surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Current then Sham then Active Current (Experimental): Electrical current will be introduced to the insulated percutaneous lead(s) for 5 minutes; then sham/placebo for 5 minutes; and then active electrical current for the following 2-4 weeks
  Interventions: Device: Percutaneous peripheral nerve stimulation; Device: Sham stimulation
- Sham then Active Current (Active Comparator): Sham/placebo will be introduced to the insulated percutaneous lead(s) for 5 minutes; then active electrical current for the following 2-4 weeks
  Interventions: Device: Percutaneous peripheral nerve stimulation; Device: Sham stimulation

INTERVENTIONS:
Device: Percutaneous peripheral nerve stimulation — Active electrical stimulation for 5 minutes in the recovery room
  Other Names: Percutaneous peripheral neuromodulation; Ultrasound-guided percutaneous peripheral nerve stimulation
Device: Sham stimulation — Sham (placebo) stimulation for 5 minutes in the recovery room
Device: Percutaneous peripheral nerve stimulation — Active electrical stimulation for 2-4 weeks at home
  Other Names: Percutaneous peripheral neuromodulation; Ultrasound-guided percutaneous peripheral nerve stimulation

SUMMARY:
The moderate-to-severe pain many patients experience following orthopedic surgery is often treated with opioids, which are associated with side effects such as nausea/vomiting, sedation, and respiratory depression (and a risk of abuse). Potent site-specific analgesia with fewer side effects may be provided with a "continuous peripheral nerve block," which involves the percutaneous insertion of a catheter adjacent to the peripheral nerve(s) supplying a surgical site. Local anesthetic is introduced via the catheter. However, there are major problems with continuous nerve blocks that have dramatically limited their use outside academic centers. Percutaneous peripheral nerve stimulation (PNS) or "nerve modulation" is an alternative method of pain control involving the insertion of an electrical lead through an introducing needle-obviating an open surgical incision for placement-followed by the introduction of electric current to produce analgesia. This modality has been used to treat chronic pain, but it has not been evaluated with a randomized, controlled study when applied to acute pain management (post-surgical analgesia). This temporary therapy has multiple theoretical benefits over existing analgesics, such as a lack of systemic side effects (e.g., nausea, respiratory depression), an absence of induced muscle weakness, and a reduced risk of adverse events (e.g. infection). The purpose of the proposed randomized, double-masked, placebo-controlled, crossover, feasibility study is to explore the possibility of treating postoperative pain with ultrasound-guided percutaneous PNS and, if so, to help power a subsequent definitive randomized, controlled trial.

DETAILED DESCRIPTION:
Written, informed consent will be obtained using an IRB-approved ICF prior to any study procedures. Lead insertion may occur up to 2 weeks prior to surgery within the CTRI, or the morning of surgery in the regional anesthesia induction area (it just depends on subject and surgeon preference, as well as logistical issues such as the time of the surgery and availability of the investigators). Muscle strength will be measured with a pressure transducer.

Preoperative lead insertion (approximately 1-3 hours). A percutaneous, helically-coiled, insulated electrical lead will be inserted via an introducer needle at least 2 cm proximal or distal to the perineural catheter location along the target nerve using real-time ultrasound guidance:

Surgical Procedure Location: Perineural Catheter Location, Electrical Lead Location

Shoulder: Interscalene, Interscalene or supraclavicular or suprascapular

At or distal to the elbow: Infraclavicular, Interscalene, supraclavicular or terminal nerve(s)

Foot or ankle: Popliteal-sciatic [adductor canal optional], Subgluteal-sciatic [femoral optional] <or vice vera>

Knee or distal thigh: Adductor canal [popliteal-sciatic optional], Femoral [subgluteal-sciatic optional]

It will be optional for a conducting probe to be used prior to lead insertion-this allows identification of the optimal lead tip location relative to the target nerve by passing electrical current via the insulated probe. The desired end point is a pleasant paresthesia in the distribution of the target nerve reported by the subject. If used, the probe will be completely withdrawn following target location identification, and a lead subsequently inserted to the target location. Following needle removal, the percutaneous helical lead will have electric current passed using the SPRINT (SPR Therapeutics, Cleveland, OH) pulse generator to ensure accurate placement (a pleasant paresthesia in the distribution of the target nerve). It will be replaced, if necessary. Muscle strength will be measured with a pressure transducer during the delivery of electrical current. The pulse generator will then be removed and the lead affixed to the skin using an occlusive dressing.

With the subject's permission the investigators may photograph or videotape the procedures described above for educational, training, or publication purposes. The photos or video will focus only on the lead insertion site and affected limb. Ultrasound images from the procedure may also be collected. Every effort will be made to protect the subject's privacy and the photos or video will not include the subject's face or any other personal identifiers such as birthmarks. Subjects and their caretakers will be trained in device care and management, and given written instructions as well. Following successful lead insertion, a perineural catheter may be inserted, if the patient desires a catheter (with normal saline injection and not local anesthetic via the inserting needle). This will be used to deliver perineural local anesthetic as a rescue analgesic method postoperatively in case the SPRINT system provides inadequate analgesia.

Randomization. Within the recovery room, the surgeon often performs a standard neurologic examination (variable depending on the surgeon and surgical procedure), after which time the subject will have baseline end points measured, including a pain score at the surgical site using the Numeric Rating Scale (NRS, 0-10), pain score (NRS) within the target nerve distribution, and sensory deficits (measured with alcohol pads and von Frey filaments compared to the contralateral limb within the cutaneous distribution of the target nerve). For their first pulse generator-"Stimulator A"-subjects will be randomized to one of two treatments-current or sham-using computer generated lists and opaque, sealed envelopes. The stimulator will then be attached to the lead and switched "on" (sham stimulator produces no current). The end points will be measured per the table below. Subsequently, the stimulator will be replaced by the alternative (current or sham)-"Stimulator B". The subject will have the end points measured and the stimulator replaced with a unit set to deliver active current for the remainder of study participation ("Stimulator C"). Operating and recovery room pharmacologic analgesic requirements will be recorded. Of note, if a lead fails to provide paresthesias within the target nerve distribution with either Stimulator A or B (adjustment of stimulator settings allowed), the lead may be replaced at the discretion of the subject and investigators.

End point collection (first day within the recovery room; approximately 30 minutes):

Baseline, then stimulator A is activated (sham or real) Minutes 1-5, then stimulator B is activated (sham or real) Minutes 1-5, then stimulator C is activated (always real) Minute 5 and 30 within the recovery room Daily x 14 days Months 1 and 3

Endpoints will include the numeric rating scale for pain (NRS) at the surgical site at rest and with movement, the lead-related NRS (pain at lead site), muscle strength, sensory deficits, and the question "adequate analgesia?" as a nominal response of yes or no.

Of note, the data derived from the chronic pain literature suggests that there is a "carry over" effect following stimulation: analgesia is provided even after the cessation of electrical current. It remains unknown if this is true following surgery in the acute postoperative pain period. For subjects randomized to active current from Stimulator A, the data collected for Stimulator B placebo treatment may be lowered due to the carry over effect. Therefore, this data will not be compared with the baseline or Stimulator A outcome measures. However, it is valuable data to possibly detect and quantify the carry-over effect of the initial stimulation.

At any time, subjects may choose to have their perineural catheter bolused with local anesthetic and a perineural local anesthetic infusion begun (if they desired a catheter with subsequent insertion). Therefore, subjects will not risk receiving inferior analgesia by participating in this study. However, subjects also have the option of leaving their infusion pump off and using neuromodulation as their primary analgesic if the latter proves adequate-the decision is completely each subject's and may be made any time prior to perineural catheter removal.

Subjects and their caretakers will be trained in device care and management, and given written instructions as well. Pain scores (resting and dynamic worst and average) will be collected daily for two weeks, along with oral analgesic requirements, perineural local anesthetic use, and sensory/motor deficits (all specific to the previous 24 hours). Perineural catheters will be removed at home upon subject request, after 3 days, or upon local anesthetic reservoir exhaustion, whichever comes first (standard-of-care). The electrical leads will be removed upon subject request, or after 30 days, whichever comes first. The leads will be removed at home by subjects or their caretakers (standard-of-care for perineural catheter withdrawal) or by investigators, depending on both investigator and subject preference. If removed by subjects or their caretakers, a picture of the extracted lead tip must be texted/emailed to investigators, or the physical lead returned to investigators for inspection. Subjects will be contacted no less than every 5 days following the initial 2-week period until their lead is removed; and, will then be contacted 1 and 3 months postoperatively and the end points again verbally collected.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing orthopedic surgical procedure that frequently results in moderate-to-severe postoperative pain
* At least 18 years of age
* Able to understand and willing to take part in study and adhere to all study requirements

Exclusion Criteria:

* Postoperative analgesic plan includes a single-injection peripheral nerve block in the surgical extremity
* Chronic opioid use (daily use within the 2 weeks prior to surgery and duration of use > 4 weeks)
* Known neuro-muscular deficit of the target nerve(s)
* Anticipated MRI within the following 2 weeks
* Compromised immune system based on medical history (e.g., immunosuppressive therapies such as chemotherapy, radiation, sepsis, infection), or other conditions that places the subject at increased risk in the opinion of the investigator
* Implanted spinal cord stimulator, cardiac pacemaker/defibrillator, deep brain stimulator, or other implantable neurostimulator whose stimulus current pathway may overlap
* History of bleeding disorder
* Antiplatelet or anticoagulation therapies other than aspirin
* Allergy to all local anesthetic agents such as lidocaine or previous reaction to anesthesia
* Allergy to skin-contact materials (occlusive dressings, bandages, tape etc.)
* Any other condition that may interfere with ability to participate in a clinical trial (e.g., anatomy that may interfere with lead placement) as determined by the Investigators
* Incarceration
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, MD, MS, Principal Investigator — University California San Diego
Locations (3):
- United States (3):
  - UCSD Medical Center, Thornton, La Jolla, California
  - Ucsd Ctri, La Jolla, California
  - UCSD Medical Center, Hillcrest, San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ilfeld BM, Gabriel RA, Said ET, Monahan AM, Sztain JF, Abramson WB, Khatibi B, Finneran JJ 4th, Jaeger PT, Schwartz AK, Ahmed SS. Ultrasound-Guided Percutaneous Peripheral Nerve Stimulation: Neuromodulation of the Sciatic Nerve for Postoperative Analgesia Following Ambulatory Foot Surgery, a Proof-of-Concept Study. Reg Anesth Pain Med. 2018 Aug;43(6):580-589. doi: 10.1097/AAP.0000000000000819. PMID 29905630
- [Derived] Ilfeld BM, Finneran JJ 4th, Gabriel RA, Said ET, Nguyen PL, Abramson WB, Khatibi B, Sztain JF, Swisher MW, Jaeger P, Covey DC, Meunier MJ, Hentzen ER, Robertson CM. Ultrasound-guided percutaneous peripheral nerve stimulation: neuromodulation of the suprascapular nerve and brachial plexus for postoperative analgesia following ambulatory rotator cuff repair. A proof-of-concept study. Reg Anesth Pain Med. 2019 Mar;44(3):310-318. doi: 10.1136/rapm-2018-100121. Epub 2019 Feb 15. PMID 30770421
- [Derived] Ilfeld BM, Said ET, Finneran JJ 4th, Sztain JF, Abramson WB, Gabriel RA, Khatibi B, Swisher MW, Jaeger P, Covey DC, Robertson CM. Ultrasound-Guided Percutaneous Peripheral Nerve Stimulation: Neuromodulation of the Femoral Nerve for Postoperative Analgesia Following Ambulatory Anterior Cruciate Ligament Reconstruction: A Proof of Concept Study. Neuromodulation. 2019 Jul;22(5):621-629. doi: 10.1111/ner.12851. Epub 2018 Aug 30. PMID 30160335

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a feasibility study and we prospectively chose a convenience sample. We decided that we had enough data from this phase after enrolling 7 subjects for the sciatic leads and therefore closed enrollment and the study.
Groups:
- Active Then Sham Then Active: electrical current will be introduced to the insulated percutaneous lead(s) for 5 minutes, then sham for 5 minutes, then active current for 2-4 weeks
- Sham Then Active Electrical Current: sham will be given for 5 minutes followed by active current for 2-4 weeks
Period: Overall Study
Arm/Group | Active Then Sham Then Active | Sham Then Active Electrical Current
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Then Sham Then Active | Sham Then Active Electrical Current | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (3.9) | 48.0 (20.8) | 55 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 0 | 1 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7
Height [Mean (Standard Deviation); unit: cm] | 163.8 (3.3) | 175.3 (19.8) | 168.7 (13.2)
Height [Mean (Standard Deviation); unit: kg] | 67.0 (10.9) | 96.8 (40.2) | 79.8 (29.2)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.0 (3.8) | 30.4 (5.2) | 27.3 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Surgical Site Pain Level (NRS) at Rest [Percentage of Baseline Pain]
Description: Pain is evaluated on a Numeric Rating Scale: 0-10 scale with 0=no pain and 10=worst imaginable pain. The outcome measure is calculated as such: the pain score 5 and then 10 minutes after the stimulator is first activated on the Numeric Rating Scale divided by the baseline pain score measured on the same scale. Of note, although this is a crossover design, the order of treatment does influence the effects of each treatment, so the 7 total subjects cannot be grouped together for the active portion and then again for the sham portion--they must remain separate, distinct groups even though this is a crossover design.
Time Frame: 5 and 10 minutes after the stimulator is first activated
Measure: Mean (Full Range); unit: percentage of baseline
Groups:
- Electrical Current: electrical current will be introduced to the insulated percutaneous lead(s) for 5 minutes
  Ultrasound-guided percutaneous peripheral nerve stimulation: Using ultrasound guidance, the small electrical lead is inserted adjacent to a target peripheral nerve through a percutaneously introduced 20-gauge needle. Following needle withdrawal, the percutaneous lead is attached to a miniature stimulator half the size of a business card that is simply adhered to the skin. When activated, the (active) stimulator generates a small electrical current which passes through the insulated leads to the uninsulated lead tip, which activates nerve fibers (placebo stimulators do not generate current).
- Placebo: NO electrical current will be introduced to the insulated percutaneous lead(s) for 5 minutes
  Ultrasound-guided percutaneous peripheral nerve stimulation: Using ultrasound guidance, the small electrical lead is inserted adjacent to a target peripheral nerve through a percutaneously introduced 20-gauge needle. Following needle withdrawal, the percutaneous lead is attached to a miniature stimulator half the size of a business card that is simply adhered to the skin. When activated, the (active) stimulator generates a small electrical current which passes through the insulated leads to the uninsulated lead tip, which activates nerve fibers (placebo stimulators do not generate current).
Arm/Group | Electrical Current | Placebo
Number analyzed (Participants) | 4 | 3
percentage of baseline
  5 Minutes after baseline just before 1st intervention | 64 [28 to 100] | 100 [100 to 100]
  10 minutes after baseline (which was just before 1st intervention) | 55 [33 to 71] | 69 [33 to 100]

2. Other Pre Specified Outcome: Percentage of Baseline Muscle Strength
Description: Strength is evaluated using an isometric force electromechanical dynamometer to measure the force produced during a maximum voluntary isometric contraction during plantar flexion. The outcome measure is calculated as such: the force produced after the stimulator is activated divided by the baseline force prior to stimulation initiation. Of note, although this is a crossover design, the order of treatment does influence the effects of each treatment, so the 7 total subjects cannot be grouped together for the active portion and then again for the sham portion--they must remain separate, distinct groups even though this is a crossover design.
Time Frame: Two minutes following stimulation initiation following lead insertion
Measure: Mean (Standard Deviation); unit: percentage of baseline muscle strength
Groups:
- Electrical Current: electrical current will be introduced to the insulated percutaneous lead for 5 minutes
- Placebo: NO electrical current will be introduced to the insulated percutaneous lead for 5 minutes
Arm/Group | Electrical Current | Placebo
Number analyzed (Participants) | 4 | 3
percentage of baseline muscle strength | 1.0 (2.1) | -2.3 (3.2)

3. Other Pre Specified Outcome: Worst Pain at Rest
Description: Pain level evaluated with a 0-10 Numeric Rating Scale with 0=no pain and 10=worst imaginable pain. Both treatment groups are receiving active stimulation from 10 minutes following baseline until the leads are removed 2-4 weeks following baseline. However, we do not know if the order of the first 10 minutes of treatment (either sham then stimulation or stimulation then sham) affects subsequent effects. Therefore, these two treatment groups must remain separate for the remainder of the study period (even though both treatment groups are receiving the same intervention on each of the days described here).
Time Frame: Daily for Days 1-14 following surgery, then at 30 and 90 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Then Sham Then Active | Sham Then Active Electrical Current
Number analyzed (Participants) | 4 | 3
score on a scale
  Day 1 following intervention | 1.7 (1.5) | 0.7 (1.2)
  Day 2 following intervention | 2.7 (2.5) | 3.0 (3.0)
  Day 3 following intervention | 1.3 (1.2) | 1.0 (1.0)
  Day 4 following intervention | 0.7 (1.2) | 0.7 (1.2)
  Day 5 following intervention | 1.3 (2.3) | 1.3 (0.6)
  Day 6 following intervention | 1.3 (2.3) | 1.0 (1.0)
  Day 7 following intervention | 2.7 (2.3) | 0.3 (0.6)
  Day 8 following intervention | 3.0 (2.6) | 0 (0)
  Day 9 following intervention | 2.3 (2.1) | 0 (0)
  Day 10 following intervention | 2.3 (2.1) | 0 (0)
  Day 11 following intervention | 3.3 (3.1) | 0 (0)
  Day 12 following intervention | 3.0 (2.6) | 0 (0)
  Day 13 following intervention | 2.3 (2.1) | 0 (0)
  Day 14 following intervention | 2.5 (2.3) | 0 (0)
  Day 30 following intervention | 0 (0) | 0 (0)
  Day 90 following intervention | 0 (0) | 0 (0)

4. Other Pre Specified Outcome: Average Pain at Rest
Description: as for outcome 3
Time Frame: Daily for days 1-14 following surgery, then at 30 and 90 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Then Sham Then Active | Sham Then Active Electrical Current
Number analyzed (Participants) | 4 | 3
score on a scale
  Day 1 following intervention | 0.5 (0.5) | 0 (0)
  Day 2 following intervention | 1.3 (1.2) | 0.7 (1.2)
  Day 3 following intervention | 1.3 (1.2) | 0.3 (0.6)
  Day 4 following intervention | 0.3 (0.6) | 0 (0)
  Day 5 following intervention | 0.3 (0.6) | 0 (0)
  Day 6 following intervention | 0.3 (0.6) | 0 (0)
  Day 7 following intervention | 0.3 (0.6) | 0 (0)
  Day 8 following intervention | 0.3 (0.6) | 0 (0)
  Day 9 following intervention | 1.0 (1.0) | 0 (0)
  Day 10 following intervention | 1.0 (1.0) | 0 (0)
  Day 11 following intervention | 1.3 (1.5) | 0 (0)
  Day 12 following intervention | 1.0 (1.0) | 0 (0)
  Day 13 following intervention | 1.0 (1.0) | 0 (0)
  Day 14 following intervention | 1.0 (1.0) | 0 (0)
  Day 30 following intervention | 0 (0) | 0 (0)
  Day 90 following intervention | 0 (0) | 0 (0)

5. Other Pre Specified Outcome: Worst Pain During Movement
Description: as for outcome 3
Time Frame: Daily for Days 1-14 following surgery, then at 30 and 90 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Then Sham Then Active | Sham Then Active Electrical Current
Number analyzed (Participants) | 4 | 3
score on a scale
  Day 1 following intervention | 2.7 (2.3) | 0.7 (1.2)
  Day 2 following intervention | 4.2 (3.7) | 2.7 (3.8)
  Day 3 following intervention | 3.0 (2.6) | 1.0 (1.0)
  Day 4 following intervention | 2.0 (2.0) | 0.7 (1.2)
  Day 5 following intervention | 2.0 (2.0) | 1.3 (0.6)
  Day 6 following intervention | 2 (2) | 1 (1)
  Day 7 following intervention | 2.7 (2.3) | 0.3 (0.6)
  Day 8 following intervention | 3.3 (3.1) | 0 (0)
  Day 9 following intervention | 2.7 (2.3) | 0 (0)
  Day 10 following intervention | 3.0 (2.6) | 0 (0)
  Day 11 following intervention | 3.7 (3.2) | 0 (0)
  Day 12 following intervention | 3.3 (2.9) | 0 (0)
  Day 13 following intervention | 3 (2.6) | 0 (0)
  Day 14 following intervention | 3 (2.6) | 0 (0)
  Day 30 following intervention | 0 (0) | 0 (0)
  Day 90 following intervention | 0 (0) | 0 (0)

6. Other Pre Specified Outcome: Average Pain During Movement
Description: as for outcome 3
Time Frame: Daily for Days 1-14 following surgery, and then at 30 and 90 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Then Sham Then Active | Sham Then Active Electrical Current
Number analyzed (Participants) | 4 | 3
score on a scale
  Day 1 following intervention | 1.2 (1.6) | 0 (0)
  Day 2 following intervention | 2 (2) | 0.7 (1.2)
  Day 3 following intervention | 2.3 (2.1) | 0.7 (1.2)
  Day 4 following intervention | 1 (1) | 0.3 (0.6)
  Day 5 following intervention | 1.2 (1.3) | 0.3 (0.6)
  Day 6 following intervention | 0.7 (1.2) | 0 (0)
  Day 7 following intervention | 1.8 (16) | 0 (0)
  Day 8 following intervention | 1.7 (1.5) | 0 (0)
  Day 9 following intervention | 1.7 (1.5) | 0 (0)
  Day 10 following intervention | 1.7 (1.5) | 0 (0)
  Day 11 following intervention | 1.8 (1.6) | 0 (0)
  Day 12 following intervention | 2 (1.7) | 0 (0)
  Day 13 following intervention | 1.3 (1.2) | 0 (0)
  Day 14 following intervention | 1.7 (1.5) | 0 (0)
  Day 30 following intervention | 0 (0) | 0 (0)
  Day 90 following intervention | 0 (0) | 0 (0)

7. Other Pre Specified Outcome: Opioid Consumption
Description: Oxycodone consumption (oxycodone is a synthetic opioid). Both treatment groups are receiving active stimulation from 10 minutes following baseline until the leads are removed 2-4 weeks following baseline. However, we do not know if the order of the first 10 minutes of treatment (either sham then stimulation or stimulation then sham) affects subsequent effects. Therefore, these two treatment groups must remain separate for the remainder of the study period (even though both treatment groups are receiving the same intervention on each of the days described here).
Time Frame: Daily for Days 1-14 following surgery, and then at 30 and 90 days
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Active Then Sham Then Active | Sham Then Active Electrical Current
Number analyzed (Participants) | 4 | 3
mg
  Day 1 following intervention | 3.3 (5.8) | 0 (0)
  Day 2 following intervention | 10 (10) | 18.3 (27.5)
  Day 3 following intervention | 0 (0) | 13.3 (23.1)
  Day 4 following intervention | 1.7 (2.9) | 5.0 (8.7)
  Day 5 following intervention | 6.7 (11.5) | 3.3 (5.8)
  Day 6 following intervention | 5 (8.7) | 0 (0)
  Day 7 following intervention | 15 (15) | 0 (0)
  Day 8 following intervention | 15 (15) | 0 (0)
  Day 9 following intervention | 8.3 (7.6) | 0 (0)
  Day 10 following intervention | 6.7 (7.6) | 0 (0)
  Day 11 following intervention | 8.3 (7.6) | 0 (0)
  Day 12 following intervention | 10 (10) | 0 (0)
  Day 13 following intervention | 8.3 (7.6) | 0 (0)
  Day 14 following intervention | 8.3 (7.6) | 0 (0)
  Day 30 following intervention | 0 (0) | 0 (0)
  Day 90 following intervention | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: 90 days
Groups:
- Stimulation: active electrical stimulation for 5 minutes followed by 5 minutes of sham and then 2-4 weeks of active electrical stimulation
- Sham: sham for 5 minutes followed by 5 minutes of active electrical stimulation and then 2-4 weeks of active electrical stimulation
Arm/Group | Stimulation | Sham
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT02898103/Prot_SAP_000.pdf